CLINICAL TRIAL: NCT00519909
Title: The Effect of Calcium on Fecal Fat and Energy Excretion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Arla Foods (Industry); The Danish Dairy Research Foundation, Denmark (Other); FOOD Graduate School, the Royal Veterinary & Agricultural University, Denmark (Other); Danish Research Agency (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H-KF-01-144/02
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Obesity
Keywords: dairy products, calcium, fat excretion, energy excretion
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Other): Diet with high content of calcium and high content of fat
  Interventions: Other: Dairy calcium
- 2 (Other): Diet with low content of calcium and high content of fat
  Interventions: Other: Dairy calcium
- 3 (Other): Diet with high content of calcium and normal content of fat
  Interventions: Other: Dairy calcium
- 4 (Other): Diet with low content of calcium and normal content of fat
  Interventions: Other: Dairy calcium
- 5 (Other): Diet with high content of calcium fra supplement and high content of fat
  Interventions: Other: Dairy calcium

INTERVENTIONS:
Other: Dairy calcium — Diets with different content of calcium and fat

SUMMARY:
The overall purpose of this study is to examine the effect of calcium on fecal fat and energy excretion.

DETAILED DESCRIPTION:
Several reports have found inverse associations between calcium intake and body weight. Few intervention studies have shown that a high calcium diet resulted in a greater body weight loss than a low calcium diet. The mechanism is not clear, but one possible explanation is reduced absorption of fat in the gut, due to formation of insoluble calcium fatty acid soaps or binding of bile acids which impairs the formation of micelles.

The aim of this study is to examined if a high calcium intake from dairy products, in diets high or normal in fat content, have an effect on fecal energy and fat excretion, concentrations of substrates involved in energy metabolism and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* healthy meals
* BMI 24-31 kg/m2
* age between 18-50 years

Exclusion Criteria:

* donation of blood 6 months before and under the study
* milk allergy, diabetes, hypertension, hyperlipidemia, cronic infectious disease
* use of dietary supplements 3 months before and under the study
* smoking
* elite athletes
* use of medication

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-08; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Fecal fat excretion, fecal energy excretion, calcium excretion, cholesterol

SECONDARY OUTCOMES:
Vitamin D, changes in lipolyse

CONTACTS AND LOCATIONS:
Overall Officials: Janne K Lorenzen, PhD student, Principal Investigator — Dept. of Human Nutrition, Faculty of Life Sciences, Univerity of Copenhagen
Locations (1):
- Dept. of Human Nutrition, Faculty of Life Sciences, University of Copenhagen, Frederiksberg, Denmark